CLINICAL TRIAL: NCT02473796
Title: Effect of Home Based Child Care on Child Mortality and Malnutrition in a Tribal Population of Melghat, India: Cluster Randomised Control Field Trial
Brief Title: Home Based Child Care to Reduce Mortality and Malnutrition in Tribal Children of Melghat, India: CRCT
Acronym: HBCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MAHAN Trust (Other)
Collaborators: Stitching Geron and Cordaid, The Netherlands. (Unknown); Caring Friends, Mumbai (Unknown)
Responsible Party: Principal Investigator, Dr. Ashish Rambhau Satav, President MAHAN Trust, MAHAN Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MT-1
Record Dates: First submitted 2015-04-10; First posted 2015-06-17 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Acute Respiratory Tract Infections; Diarrhea; Malaria; Neonatal Sepsis; Birth Asphyxia
Keywords: home based child care
MeSH Terms: conditions — Diarrhea; Malaria; Neonatal Sepsis; Asphyxia Neonatorum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home based child care (Experimental): The home based child care included treatment of various various childhood illnessed by locally avialable trained village health workers, improving hygiene and nutrition among children and women throgh health education. This care was in adiition to the local health care provided by the Government's primary health care services.
  Interventions: Other: Home based child care
- control (No Intervention): The control arm included population where the home based neonatal care was not implimented. The health services were provided by the Government run primary health care services. Vital statistics data was collected by VHWs.

INTERVENTIONS:
Other: Home based child care — HBNC included treatment of neonatal sepsis with Gentamicin once daily (5 mg for 10 days for preterm babies with birth weight <2000g; 7 mg for birth weight 2000-2500 gm or as per gentamicin chart for 7 days for normal term & weight ) by intramuscular injection. Acute respiratory infection was treated with co-trimoxazole syrup BID (2.5 ml for age 1-2 months, 5 ml for age 2 months - 1 year, 7.5 ml for age 1 - 5 years). Diarrheal illness was treated with ORS, furoxone (5 ml 8 hourly for 3 days) and metronidazole syrup (5 ml 8 hourly for 7 days). Malaria was treated with Syrup chloroquine (for 1 month to 1 year- 5 ml first dose , 2.5 ml after 6 hours, 2.5 ml after 12 hours , 2.5 ml after 12 hours). Syrup paracetamol was given 2.5 to 5 ml 8 hourly depending upon the body weight.
  Other Names: HBCC
  Arms: Home based child care

SUMMARY:
Melghat is poorly developed tribal area in India with very high child mortality & malnutrition prevalence (grossly inadequate medical facilities). Important health problems. Malnutrition , Pneumonia, Tuberculosis, Anaemia, Malaria, Diarrhoea, Premature and L. B. W. babies, Neonatal sepsis, Feeding problem, Birth asphyxia. The investigators developed a Home Based Child Care (HBCC) model to reduce neonatal mortality rate (NMR), infant mortality rate (IMR), under 5 mortality rate (U5MR) and severe malnutrition(SM) in this region.

Melghat.

Need of project :

Melghat is known for highest U5MR in Maharashtra. Overall aims and importance of the research:. The results obtained in this area will be applicable for reducing children mortality and malnutrition in other parts of Melghat and all other tribal areas of India.

Methodology: RCT-Home based child care (HBCC) by trained village health workers .(ARI, Diarrhoea, Malaria clinically & Neonatal care) in 19 villages. Strengthening of existing government ICDS and health system.

Melghat.

Need of project :

Melghat is known for highest U5MR in Maharashtra. Overall aims and importance of the research:. The results obtained in this area will be applicable for reducing children mortality and malnutrition in other parts of Melghat and all other tribal areas of India.

Methodology: RCT- (HBCC) by trained village health workers .(ARI, Diarrhoea, Malaria clinically & Neonatal care) in 19 villages.

DETAILED DESCRIPTION:
A. Objectives:

1. To reduce NMR from existing 54 ( year 2004) to 33.6 per 1000 live births in usual residents population of 17000 (from 19 villages in tribal area of Melghat ) over a period of 5 years.
2. To reduce the IMR from existing 90 (year 2004) to 52.65 per 1000 live births in above area.
3. To reduce the U5MR from existing 140 (year 2006) to 72.1 per 1000 live births in above area.
4. To reduce the prevalence of severe malnutrition (under 5 children ) from existing 9.5% (year 2004) to 4.55% in above area.

B. Detailed research plan. I. Study design: Randomised Control Trial. The Melghat area was divided into 5 clusters. 8 villages were randomly selected from each cluster by lottery method. All under 5 children who are ill will be treated by trained VHW.

II. Study period: January 1st, 2004 to 31st April, 2010. III. Study area: 19 villages for intervention and control area with Population of 14888 & 16310 respectively.

IV) Contents of the home based child health Package:

A. Provision of home based health care. It comprises provision of home-based health care to pregnant mothers and under 5 children through a trained semi-literate female village health worker (VHW) resident of the same village under medical supervision by trained medical supervisor.

Arms Experimental: Home based child care The home based child care included treatment of various childhood illnesses by VHWs, improving hygiene and nutrition among children and women through health education.

Assigned interventions Home based child care Other Names: HBCC included treatment of neonatal sepsis with Gentamicin once daily (5 mg for 10 days for preterm babies with birth weight <2000g; 7 mg for birth weight 2000-2500 gm or as per gentamicin chart for 7 days for normal term & weight ) by intramuscular injection.

Acute respiratory infection was treated with co-trimoxazole syrup BID (2.5 ml for age 1-2 months, 5 ml for age 2 months - 1 year, 7.5 ml for age 1 - 5 years).

Diarrheal illness was treated with ORS, furoxone (5 ml 8 hourly for 3 days) and metronidazole syrup (5 ml 8 hourly for 7 days).

Malaria was treated with Syrup chloroquine (for 1 month to 1 year- 5 ml first dose , 2.5 ml after 6 hours, 2.5 ml after 12 hours , 2.5 ml after 12 hours). Syrup paracetamol was given 2.5 to 5 ml 8 hourly depending upon the body weight.

Placebo Comparator: control The control arm included population where the HBCC was not implemented.

Both arms: The health services were provided by the Government run primary health care services. Vital statistics data was collected by VHWs.

D) Studies of prevalent knowledge and attitudes of the community regarding maternal and child health .

V) The team of workers under the program are as follows:

i) VHW: 19 Trainer and guide of the VHWs: ii) 2 medical supervisors, iii) 2 nutrition supervisors iv) 2 vital statistic supervisors.

v) The Traditional Birth Attendant (TBA). vi) A project manager. vii) One doctor will guide, train, examine neonates (1st day) and evaluate the program.

VI. Implementation of HBCC

HBCC is a community-based project and following are the main components:

Micro plan preparation includes following:

i) Objectives, activities and methods. ii) Area & socio-economic profile. iii) Map of the area. iv) Distribution and allocation of villages to VHW: v) Clear definitions of roles and responsibilities of workers. vi) GANTT chart vii) VHW's emolument or earning. viii) Check-list for supervisor & VHW activities. x) Community involvement xi) Budget xii) KAP of traditional care. xiii) TBAs involvement xiv) Placement of the supervisor VII.

1. The total duration of training for supervisors and VHWs is 45 days. 2. TBAs are trained in three workshops each of two-day duration.

VIII. Collection of Vital Statistics: VHWs will collect death and birth records. The vital statistics supervisor will supervise it. Retrospective surveyor will conduct house-to-house survey every six months to collect these data independently. TBAs will assist.

IX. Monitoring & Evaluation of project:

Monitoring indicators for the objective:

Monitor monthly: No. of pregnant ladies, VHW attendance during deliveries, No. of neonates started breast feeding within 60 min, No. of patients treated, etc.

Evaluation of project:

A. External evaluation. B. Outcome evaluation - Mortality and morbidity (malnutrition ) will be measured and reported in the outcome measure tables .

i ) NMR, IMR, CMR, ( children deaths per 1000 live births) ii) Prevalence of severe malnutrition(SM). (percentage of children) The secondary outcome measure, prevalence of SM was determined by weight of child in Kilogram versus age of child in months, in September of each year. Indian Academy of Paediatrics classification was used for gradation of malnutrition. Gr. III and IV =Severe malnutrition. Weight of child will be measured and reported.

C. Process evaluation. Data analysis by Microsoft Excel and fox pro.

X. Phases: Three distinct phases are:

1. The first year of training, Observation, baseline data collection and recording.
2. Post-neonatal disease management from May 2005.
3. Providing HBCC services from May 2005 to April 2010. Data analysis from May 2010 to July 2010.

XI. The physical inputs Items in the VHW Kit Wrist Watch, digital thermometer, Salter weighing Scale. Adult weighing scale, Ambu bag, Warm bag , Blankets, Kangaroo mother care blouse, Mucus extractor, Health education flipchart , Special spoon for feeding neonates, etc. Tab Paracetamol 500 mg, Gentian violet paint 400 ml bottle, Injection Gentamicin vial 2 ml vial ( 40 mg per ml), Surgical cotton, Tab. Co- trimoxazole-Trimethoprim 20 mg +Sulphamethoxazole 100 mg, Syrup Co- trimoxazole-Trimethoprim 40 mg +Sulphamethoxazole 200 mg , Spirit, Insulin Syringe, Tab Salbutamol- 2mg , Injection Vitamin K 10 mg ampoule. Chloromycetin eye applicap. Oral Rehydration solution. Tab. Albendazole, Syrup Chloroquine , Tab. Furoxone, Syrup Furoxone, Syrup Metronidazole, Syrup Albendazole, Syrup Paracetamol, Tab. Domperidone 5 mg, Tab. CPM. Antiseptic powder (10gram), Adhesive plaster, etc.

XII. Facilities available at the sponsoring institution:

Two full time well experienced post graduate doctors , trained VHWs(19), medical supervisors (2) and project director. Facilities for hospitalization and training of VHWs.

XIII. Total Budget (costs)- The cost of implementation of HBCC may be around Rs.5646620 for 3 years. i. Staff: 2323850 ii. Contingencies 16000 Recurring: 3774999 Total Non-recurring: 1602725 iii. Audit & Administration: 268896.22

Annexure:

1. Activities under HBCC: Treatment of under 5 children, normal neonatal care , growth monitoring & vital statistics data collection by VHWs in the intervention villages will be a regular activity. Retrospective survey and data analysis of IA & CA will be conducted every 6 months.

Periodic activities are: Gramsabha, Program manager, project director village visit, Launch, BCC- community or group health education, Counting of under 5 children once a year, Training of VHW and supervisors, Weight record of under 5 children in intervention area, Midterm evaluation, final data analysis and final evaluation by external agencies.

Annexure 2- Socioeconomic profile of intervention area. Melghat is hilly forest area with 317 villages in central India . Population is 2,50,000 & 75% of them are tribal . Most of the tribal(>90 %) are farmers or labourers living very hard life, below poverty line(>75%) & illiterate (>50%), living in huts(>90%).

Medical facilities are grossly inadequate. Annexure 3: Clear definitions of roles and responsibilities of categories of workers.

The traditional birth attendant ( TBA)

1. Reinforce the health education messages given by VHWs to pregnant mothers and her relatives.
2. Encourage mother to access ANC from the regular government health services.
3. Conduct hygienic and safe delivery.
4. Recognize danger signals in mother ( delivery, post-partum) and refer.
5. Insist that family calls VHW to assist her during delivery & work in collaboration with VHW.

The village health worker (VHW): Job description under HBCC:

VHW is the direct provider of components of the HBCC. Record keeping of the target group and work in smooth collaboration with TBA. Periodically visit every house and collect information related to pregnancy and child health.

Refer pregnant women to ANM for iron, folic acid & tetanus toxoid injection. Organize and assist supervisors in conducting group health education for pregnant women.

Make three antenatal visits to pregnant women in the village at 4th, 7th and 9th month of pregnancy for health screening, health education, Danger signs in pregnancy, labour & action to be taken. Planning for delivery & Breast feeding.

Attend delivery and observe baby

a. Record information on delivery and birth . b. Encourage cleanliness. c. Observe the new-born baby at 30 seconds after birth for cry, respiration and movement of limbs.

d. Determine whether the baby is normal or asphyxiated or still birth: and if the baby is not normal initiate asphyxia management.

g. Dry and wrap the baby h. Initiate breast-feeding. Provide care for the normal new-born . Provide care for the high risk new-born. Give Vitamin K injection. Conduct 7 regular home visits.

Identify and manage following problems in mother and new-born baby Asphyxia, Premature birth, Low birth weight, Hypothermia, Breast feeding problem, Neonatal sepsis & Pneumonia. Refer to hospital if no response in 24 hours.

Provide treatment to children of 1 months to 5 years and fill the forms for a. Pneumonia, b. Diarrhoea and dysentery, c. Malaria. d. Management of malnutrition.

3) The trainer cum medical supervisor of the VHWs. The supervisor of the VHWs is responsible for training of the VHWs in classrooms and on-going training in the field during supervisory visits, providing support and guidance to the VHWs in their work.

Job Description :

I. Checking of medicine, equipments, forms , etc. II. Visit each new-born twice. III. Supply medicines to VHW. IV. Examination of resistant malnourished cases. V. Conduct meeting of pregnant women for Health Education. VI. Proper medicine stock record. VII. Visit to patients treated by VHW. VIII. ANC B.P. record. IX. Monitoring immunization status.

4. Nutrition supervisor

1. Cross check 25% of all weights.
2. Preparation of Growth Chart & Grading of children.
3. Selection and enrolment of children & mothers for supplementary feeding.
4. Check the efficiency of weighing machine.
5. Health Education on nutrition .
6. Training & monitoring of VHW activities.
7. Arrange paediatrician visit to non-responding malnourished cases.
8. Survey of nutrition status & local food materials.
9. Motivation of people for use of local nutritious food material.
10. Identify specific nutrition deficiencies e.g. vitamin A deficiency.
11. Supply growth cards to PEM children. 5) The Project Manager The project manager has to shoulder the responsibility of ensuring that the HBCC is provided properly and that the desired outcome of reduction in mortality rates is achieved. Besides planning, resource management, overseeing execution, monitoring and evaluation of the implementation of the HBCC approach from time to time, specifically he has to undertake following responsibilities.

    1. Maintaining rapport with the community.
    2. Making available existing infrastructure.
    3. Recruitment and deployment of staff.
    4. Organizing training.
    5. Gathering data and its analysis through a competent organization.
    6. Network management etc.
    7. Ensuring availability of material.
    8. Financial monitoring,
    9. Preparing reports. Annexure :4 -Community Involvement including awareness, consent and acceptance.

Community participation may be sought at the following stages:

Key person visits, Village meetings, The village should be invited to recommend potential candidates for the work of VHWs, Launch meetings, Periodic interactions with the village to give feedback and encourage suggestions, women's micro-credit groups , Village health committee & Village Councils, etc

ELIGIBILITY:
Inclusion Criteria:

* All births and deaths in the village or catering hospital were included in the study.
* All under 5 children in the villages were included in the study.

Exclusion Criteria:

* All births and deaths outside the village were excluded from the study.

Ages: 1 Minute to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7594 (Actual)
Dates: Start 2004-01; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Under-5 mortality rate | Four years.

SECONDARY OUTCOMES:
prevalence of severe malnutrition | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ashish R Satav, MBBS., MD., Principal Investigator — MAHAN
Locations (1):
- MAHAN Trust, Melghat (Dharni), Amravati, Maharashtra, India

REFERENCES:
- [Derived] Satav AR, Satav KA, Bharadwaj A, Pendharkar J, Dani V, Ughade S, Raje D, Simoes EAF. Effect of home-based childcare on childhood mortality in rural Maharashtra, India: a cluster randomised controlled trial. BMJ Glob Health. 2022 Jul;7(7):e008909. doi: 10.1136/bmjgh-2022-008909. PMID 35851283